CLINICAL TRIAL: NCT05483946
Title: Validation of CPM#1 Compressibility Ratio in a Clinical Study of Healthy Volunteers: Evaluation of the Test-retest Repeatability
Brief Title: SWISS_CLEARANCE - Compartment Compressibility Monitoring Using CPM#1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Compremium AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SWISS_CLEARANCE
Record Dates: First submitted 2022-07-28; First posted 2022-08-02 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Compartment Syndromes
MeSH Terms: conditions — Compartment Syndromes

STUDY DESIGN:
Masking Description: Investigators will be blinded to the measurement results
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CPM#1 (Experimental): Compartment compressibility ratio measurement using the CPM#1 device
  Interventions: Device: Measurement of compartment compressibility

INTERVENTIONS:
Device: Measurement of compartment compressibility — Application of the CPM#1 device for compartment compressibility ratio measurement - for each participant, a pre-defined number of measurements will be conducted per leg and forearm

SUMMARY:
Compartment syndrome is a very serious musculoskeletal disorder, which can lead to potentially devastating consequences, such as limb amputation and life- threatening conditions. It is a well described medical condition considered to be an orthopaedic emergency affecting all ages.

Even though compartment syndrome is a well described medical condition, the appropriate treatment (i.e., fasciotomy to release tissue pressure) is invasive and involves its own risks. Furthermore, and of most critical importance is the timing for the intervention of a fasciotomy. The concerned limb may already have had severe, sometimes even irreversible, tissue damage due to high intra- compartmental pressure within 6 to 10 hours.

The standard diagnostic method for compartment syndrome is an invasive intra-compartmental pressure measurement via insertion of a pressure monitoring device into the muscle compartment. Commercially available intra compartmental pressure monitors have a highly variable intra-observer reproducibility and user errors are common.

Compared to the invasive modalities, the Compremium Compartmental Compressibility Monitoring System (CPM#1) shows promising advantages for the clinical application. Not only is the technology used for the CPM#1 device safe and non-invasive for the patient with only initial training required for the healthcare professionals, but it has also demonstrated high intra- and inter- observer reproducibility (as per bench tests and clinical settings with prototypes, to be confirmed in clinical studies like this one). The use of the CPM#1 device therefore facilitates the measurements, as it is based on pre-existing ultrasound methods and avoids any further risks to the patients compared to invasive compartmental pressure diagnosis methods.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer
* Male or female
* Age 18 to 84 years

Exclusion Criteria:

* Previous surgery to or fracture of the leg and/or forearm
* Peripheral arterial or venous disease
* History of compartment syndrome
* Limb anomalies
* General muscle disorder

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Inter-operator reproducibility with 3 raters | During the procedure which should last about 3 hours/patient
  Inter-operator reproducibility will be assessed using intra-class correlation coefficients (two-way random effects, single rater, absolute agreement). Three independent raters will conduct 4 measurements per compartment site on 14 relaxed forearms (7 volunteers, 1 site per forearm), and 14 relaxed legs (7 volunteers, 2 sites per leg).

SECONDARY OUTCOMES:
Intra-operator reproducibility | During the procedure which should last about 3 hours/patient
  Intra-operator reproducibility will be assessed using intra-class correlation coefficients (two-way mixed effects, single measurement, absolute agreement). Three independent raters will conduct 4 measurements per compartment site on 14 relaxed forearms (7 volunteers, 1 site per forearm), and 14 relaxed legs (7 volunteers, 2 sites per leg).
Validation of number of measurement repetitions | During the procedure which should last about 3 hours/patient
  Clinically needed number of measurements for optimized repeatability will be assessed on 2, 3 and 4 measurement repetitions per compartment site based on 14 relaxed forearms (7 volunteers, 1 site per forearm), and 14 relaxed legs (7 volunteers, 2 sites per leg).

OTHER OUTCOMES:
Assessment of adverse events and serious adverse events | During the procedure which should last about 3 hours/patient
  Safety of the procedure will be assessed by documenting adverse events and serious adverse events (description of the adverse events, number of participants).
Assessment of device deficiencies | During the procedure which should last about 3 hours/patient
  Safety of the procedure will be assessed by documenting device deficiencies (description)

CONTACTS AND LOCATIONS:
Overall Officials: Beat Lehmann, Principal Investigator — Universitäres Notfallzentrum, Inselspital Bern
Locations (1):
- Universitäres Notfallzentrum, Inselspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No